CLINICAL TRIAL: NCT05840328
Title: INTRAVENOUS Versus EPIDURAL DEXMEDETOMIDINE for ANALGESIA in NORMAL VAGINAL DELIVERY: A RANDOMIZED CONTROLED STUDY
Brief Title: DEXMEDETOMIDINE in NORMAL VAGINAL DELIVERY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11/2022ANET49
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Painless Vainal Labour
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- plan group (Placebo Comparator): bupivacaine will be administered epidurally as a loading dose then epidural continuous infusion with 0.125 % bupivacaine at rate 10 ml will be a maintainance for analgesia .IV placebo (normal saline) infusion will be connected to each patient at a rate of 10 ml \hr.
  Interventions: Drug: Bupivacaine Injection
- epidural group (Active Comparator): 10 ml of 0.125 % buoivacaine with 0.5 µg\ml dexmetomidine as a loading dose then continuous epidural infusion of 0.125% bupivacaine with 0.5µ/ml dexmetomidine at a rate of 10 ml\hr will be used as maintainance . IV placebo (normal saline) infusion will be connected to each patient at a rate of 10 ml\hr
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Bupivacaine Injection
- intravenous group (Active Comparator): continuous intravenous dexmetomidine infusion at rate of 0.5 µg / kg / hour in addition to same epidural infusion of 0.125% bupivacaine
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — interventional drug will be administred either intravenously or epidurally
  Arms: epidural group; intravenous group
Drug: Bupivacaine Injection — intervention drug will be administred epidurally

SUMMARY:
compare the effect of intravenous and epidural dexmetomidine as an adjuvant to local anesthetics in epidural labor analgesia in normal labor

ELIGIBILITY:
Inclusion Criteria:

* Full term (≥ 37 weeks) healthy primigravida parturients ASA2
* with single fetus scheduled for vaginal delivery
* with cephalic presentation
* requesting labor analgesia.

Exclusion Criteria:

* Allergy to dexmetomidine.(based on previous history)
* Cardiac conduction abnormalities.(all degrees of heart block , tachyarrythmias)
* Twins.
* Malpresentation.
* Preeclampsia or gestational hypertension
* Uncontrolled diabetes HBA1c ≥ 6.5%
* Uncontrolled renal failure
* Uncontrolled liver disease
* Bleeding tendency or coagulopathy.
* Contraindication or patient refusal to epidural block.
* Body mass index ≥ 35.

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-06-05 (Estimated); Study Completion 2023-07-05 (Estimated)

PRIMARY OUTCOMES:
pain relief | at 30 min after induction of block
  VAS score from 0 to 10 will be assesed
pain relief | on delivery
  VAS score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: mostafa M mansour, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No